CLINICAL TRIAL: NCT04360733
Title: Precision Immunology Approach to Better Understand the Divergent Host Responses Towards Infection With SARS-CoV-2
Brief Title: Precision Immunology to Determine the Immune Response in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bonn (Other)
Responsible Party: Principal Investigator, Dr. Christian Bode, Principle Investigator, University of Bonn
Other Study IDs: BOST-03
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV 2; COVID
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood including Serum and Immune cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- asymptomatic Covid-19: Patients with confirmed SARS-CoV2 PCR but no clinical symptoms
  Interventions: Other: Blood draw
- symptomatic Covid-19: Patients with confirmed SARS-CoV2 PCR and light clinical symptoms
  Interventions: Other: Blood draw
- severe Covid-19: Patients with confirmed SARS-CoV2 PCR and severe clinical symptoms with ICU admission
  Interventions: Other: Blood draw
- healthy controls: Persons with negative SARS-CoV2 PCR
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw — serial blood draw and subsequent deep immune phenotyping analysis, (ii.) immune activation assays, (iii.) transcriptome and (iv.) epigenome analysis in an overarching (v.) bioinformatics data analysis

SUMMARY:
To better understand the immune response to SARS-CoV-2 infection, we devised a precision immunology approach to systematically study the immune function of different patient cohorts

ELIGIBILITY:
Inclusion Criteria:

* SARS-Cov2 positive PCR

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with different severity of COVID-19. From asymptomatic to critical illness
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Immune response | 4 weeks
  Immune response of whole blood stimulation assay with various immune activators will be measured by FACS and multiplex Assay

CONTACTS AND LOCATIONS:
Overall Officials: Eicke Latz, Prof, Study Director — Institute of Innate Immunity, Univeristy of Bonn
Locations (1):
- University Hospital Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided